CLINICAL TRIAL: NCT06530030
Title: Prospective, Observational Study of the Impact of Efanesoctocog Alfa (ALTUVIIIO®) on Goal Attainment and Physical Activity in People With Moderate or Severe Hemophilia A
Brief Title: Goal Attainment and Physical Activity in People With Hemophilia A
Acronym: ACTIVIIITY
Status: Terminated | Type: Observational
Why Stopped: Early discontinuation based on sponsor decision not driven by any safety concerns.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18140; U1111-1306-7241 (Other: WHO ICTRP)
Record Dates: First submitted 2024-07-17; First posted 2024-07-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | US Export: No

GROUPS / COHORTS (1):
- Cohort: patients aged 12 to 50 years with moderate or severe hemophilia A who are newly starting prophylaxis with efa
  Interventions: Drug: efanesoctocog alfa

INTERVENTIONS:
Drug: efanesoctocog alfa — All treatment decisions must be made independent of study participation and study-related visits/assessments are not intended to inform treatment decisions. No study medication is provided as part of study participation.
  Other Names: Altuviiio

SUMMARY:
This is a Phase 4, multi-center, observational study conducted in patients aged 12 to 50 years with moderate or severe hemophilia A who are newly starting prophylaxis with efa in the US and Japan.

This study aims to enroll 35 patients.

ELIGIBILITY:
Inclusion Criteria:

* At enrollment, newly starting prophylaxis therapy with efanesoctocog alfa according to usual clinical practice, with efanesoctocog alfa initiated within 6 months after the enrollment visit
* Diagnosis of moderate (endogenous FVIII activity between 1% to 5% of normal) or severe (endogenous FVIII activity <1% of normal) hemophilia A
* Aged 12 to 50 years at time of enrollment, inclusive
* Access to a smartphone device (Android version 12.0 or higher; or iOS 13 or higher) with Bluetooth 4.0 (minimum) or 5.0 (recommended) capabilities for compatibility with physical activity tracker
* Availability of home-based access to internet for electronic patient-reported outcome (ePRO)/diary assessments
* Willingness to utilize the activity tracking device

Exclusion Criteria:

* Current diagnosis of a FVIII inhibitor, defined as inhibitor titer ≥ 0.60 BU/mL
* Use of efanesoctocog alfa for prophylaxis in the 6 months prior to enrollment

NOTE: Other Inclusion/Exclusion criteria may apply. The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with moderate or severe Hemophilia A
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Proportion of total goals achieved | Month 3
  Reported as number of individual goals with a raw GAS score of 0, +1, or +2 divided by the total number of goals set
Proportion of total goals achieved | Month 6
Proportion of total goals achieved | Month 9
Proportion of total goals achieved | Month 12
Proportion of patients who reached a +2 or +1 on at least one goal | Month 3
  Each goal will be ranked in a 5-point Likert scale ranging from +2 to -2 with +2 indicating a better goal achievement.
Proportion of patients who reached a +2 or +1 on at least one goal | Month 6
Proportion of patients who reached a +2 or +1 on at least one goal | Month 9
Proportion of patients who reached a +2 or +1 on at least one goal | Month 12
Overall GAS score | Month 3
  Goal Attainment Scaling (GAS) is a patient-centric clinician-reported outcome measure utilized to select and scale goals, with higher scores indicating greater goal attainment.
  An overall GAS score utilizing all goals set by a patient at each time point of interest will be calculated.
Overall GAS score | Month 6
  Goal Attainment Scaling (GAS) is a patient-centric clinician-reported outcome measure utilized to select and scale goals, with higher scores indicating greater goal attainment.
  An overall GAS score utilizing all goals set by a patient at each time point of interest will be calculated.
Overall GAS score | Month 9
  Goal Attainment Scaling (GAS) is a patient-centric clinician-reported outcome measure utilized to select and scale goals, with higher scores indicating greater goal attainment.
  An overall GAS score utilizing all goals set by a patient at each time point of interest will be calculated.
Overall GAS score | Month 12
  Goal Attainment Scaling (GAS) is a patient-centric clinician-reported outcome measure utilized to select and scale goals, with higher scores indicating greater goal attainment.
  An overall GAS score utilizing all goals set by a patient at each time point of interest will be calculated.
Frequency of selection of category of physical activity | Baseline
  Categories of the goals selected from the goal inventory
Monthly average of daily step count | From Baseline to Month 12
  The monthly average of daily step count (recorded by physical tracker) will be calculated using the total steps recorded in a 30-day period, accounting for the number of compliant days in that period.
Monthly average of daily activity count | From Baseline to Month 12
  Activity count includes: time spent in x, y, and z axes, vector magnitude counts, estimated calories, wear time, time spent in locomotion and non-locomotion. Counts will be averaged across the month.
Monthly average of daily Metabolic equivalent of tasks (MET) | From Baseline to Month 12
  Estimated by the physical activity tracker
Monthly average of daily Moderate and Vigorous Physical Activity (MVPA) | From Baseline to Month 12
  Summarized from MET data with time spent in moderate intensity, and vigorous intensity physical activity
Monthly average of daily intensity gradient | From Baseline to Month 12
  The intensity gradient is a measure of activity intensity distribution that reflects the distribution of intensity of physical activity by modeling the relationship between intensity and time.
Monthly average of weekly intensity gradient | From Baseline to Month 12

SECONDARY OUTCOMES:
Change in PROMIS Pain intensity score | From Baseline to Month 12
  Patient-Reported Outcome Measurement Information System (PROMIS): assessment of pain over the prior 7-day period (2 of the 3 questions) and right now (1 of the 3 questions), with patients rating their pain on a scale of 0 (had no pain) to 5 (very severe). Total score ranges from 0 to 15 and a higher score indicates worst pain intensity.
Change in HAL Score | From Baseline to Month 12
  Hemophilia Activities List (HAL) is a 42-item questionnaire to access patient ability across 7 domains: lying down/ sitting/ kneeling/ standing (8 items), functions of the legs (9 items), functions of the arms (4 items), use of transportation (3 items), self-care (5 items), household tasks (6 items), and leisure activities (7 items). Patients rate each question on a Likert scale ranging from 1 (impossible) to 6 (never). Several items have a "not applicable" option as well. There is also a visual analog scale allowing patients to self-report an overall score. A normalized total score (sum of all normalized domains) ranges from 0 (the worst possible functional status) to 100 (the best possible functional status)
Change in PROMIS pediatric Pain intensity score | From Baseline to Month 12
  Assessment of the average pain over the prior 7-day period, with patients rating their pain on a scale of 0 (no pain) to 10 (worst pain they can think of). A higher score indicates worst pain intensity.
Change in PedHAL Score | From Baseline to Month 12
  Pediatric Hemophilia Activities List (PedHAL) is a 53-item questionnaire to access patient functional ability across 7 domains: lying down/ sitting/ kneeling/ standing (10 items), functions of the legs (11 items), functions of the arms (6 items), use of transportation (3 items), self-care (9 items), household tasks (3 items), and leisure activities and sports (11 items). Patients rate each question on a Likert scale ranging from 1 (impossible) to 6 (never). Several items have a "not applicable" option as well. There is also a visual analog scale allowing patients to self-report an overall score. A normalized total score (sum of all normalized domains) ranges from 0 (the worst possible functional status) to 100 (the best possible functional status).
Change in school/work hours missed as assessed by WPAI+CIQ:HS | From Baseline to Month 12
  The Work Productivity and Activity Impairment plus Classroom Impairment Questions: Hemophilia Specific (WPAI + CIQ: HS) is a 9-item questionnaire assessing the effect of hemophilia on patients' ability to work and/or attend classes.
Change in productivity as assessed by WPAI+CIQ:HS | From Baseline to Month 12
  The Work Productivity and Activity Impairment plus Classroom Impairment Questions: Hemophilia Specific (WPAI + CIQ: HS) is a 9-item questionnaire assessing the effect of hemophilia on patients' ability to perform regular daily activities.
Change in impact on other activities as assessed by WPAI+CIQ:HS | From Baseline to 12 months
  The Work Productivity and Activity Impairment plus Classroom Impairment Questions: Hemophilia Specific (WPAI + CIQ: HS) is a 9-item questionnaire assessing the effect of hemophilia on patients' ability to perform other activities.
Mean change in total and joint domain scores of HJHS | From Baseline to 12 months
  The Hemophilia Joint Health Score (HJHS) assesses 6 index joints (left and right elbows, knees and ankles) and a global gait. For each of the 6 joints, the following items are scored: swelling (scored 0-3), duration of swelling (0-1), muscle atrophy (0-2), crepitus on motion (0-2), flexion loss (0-3), extension loss (0-3), joint pain (0-2), and strength (0-4). The HJHS provides a total score (0-124 points with higher score indicating worse joint health), joint specific scores (0-20 points), and a global gait score (0-4 points).
Monthly total and average of daily time spent in different intensity levels | From Baseline to Month 12
  Physical activity intensity defined as sedentary behavior, light intensity, moderate intensity, and vigorous intensity,
Monthly average of daily median activity count overall among moderate activities and among vigorous activities | From Baseline to Month 12
  Daily median time spent in moderate and vigorous physical activity will be averaged across the month
Monthly average of daily median MET overall among moderate activities and among vigorous activities | From Baseline to Month 12
Monthly average of weekly power law exponent alpha | From Baseline to Month 12
Monthly average of median bout length and percent of time of bout length > median bout length for each intensity level | From Baseline to Month 12
Monthly average of weekly 80th, 90th, 95th, and 100th percentiles of activity count | From Baseline to Month 12
Monthly average of weekly 80th, 90th, 95th, and 100th percentiles of MET | From Baseline to Month 12
Monthly total step count | From Baseline to Month 12
Monthly total activity count | From Baseline to Month 12
  Activity count includes: time spent in x, y, and z axes, vector magnitude counts, estimated calories, wear time, time spent in locomotion and non-locomotion. Counts will be totaled across the month.
Monthly total MET | From Baseline to Month 12
Monthly total moderate or vigorous physical activity (MVPA) | From Baseline to Month 12
  Time spent in MVPA will be totaled across the month.
Weekly average of daily step count | From Baseline to Month 12
Weekly average of daily activity count | From Baseline to Month 12
  Activity count includes: time spent in x, y, and z axes, vector magnitude counts, estimated calories, wear time, time spent in locomotion and non-locomotion. Counts will be averaged across the week.
Weekly average of daily MET | From Baseline to Month 12
Weekly average of daily MVPA | From Baseline to Month 12
  Time spent in MVPA will be averaged across the week.
Weekly average of daily intensity gradient | From Baseline to Month 12
Weekly intensity gradient | From Baseline to Month 12
Number of participants with AE, SAEs, AESIs | Baseline to end of study (12 months)
Number of participants with AEs, SAEs, AESIs related to efanesoctocog alfa | Baseline to end of study (12 months)
Proportion of total planned doses that were missed | From baseline to end of study (12 months)
Average time between treatment dose and physical activity | From baseline to end of study (12 months)
Number of patients with no reported bleeds requiring treatment | From baseline to end of study (12 months)
Average number of per patient treatment doses administered for treatment of bleeds | From baseline to end of study (12 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Bleeding and Clotting Disorders Institute, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org